CLINICAL TRIAL: NCT07312968
Title: AI4Triage - Development of an Artificial Intelligence Based Methods for the Analysis of Triage Data
Status: Active, not recruiting | Type: Observational
Sponsor: University of Catanzaro (Other)
Collaborators: Azienda Ospedaliero Universitaria Renato Dulbecco (Unknown)
Responsible Party: Principal Investigator, Pietro Hiram Guzzi, Full Professor, University of Catanzaro
Other Study IDs: AI4Triage
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Triage
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — there is no intervetiuons

SUMMARY:
Artificial intelligence, and in particular Graph Neural Networks (GNNs), have shown enormous potential in the analysis of complex clinical data. Thanks to their ability to model relationships between variables, GNNs represent a significant evolution compared to traditional models, enabling better interpretation of medical information and supporting data-driven decision-making in complex contexts such as emergency medicine.

The application of GNNs to clinical triage and to the prediction of length of stay can improve clinical efficiency by optimizing resource allocation and patient management. This observational study aims to evaluate the accuracy of predictions with respect to real clinical data, contributing to the development of advanced predictive tools to support healthcare decision-making processes.

ELIGIBILITY:
Inclusion Criteria:

* all

Exclusion Criteria:

* Patients labelled with red codes and serious injuries.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals who request access to the ER will be duly considered.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of Undertriaged | 12 monthds
  The investigators will measure the number of misclassifications
Undertriaged | 12 months
  The investigators will measure the ability to predict undertriage

CONTACTS AND LOCATIONS:
Locations (1):
- University of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Undecided